CLINICAL TRIAL: NCT02567942
Title: Assessment of the Anesthetic Effect on the Activity of Immune Cell in Patient With Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KUH1160089
Record Dates: First submitted 2015-09-02; First posted 2015-10-05 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol group (Other): The patient who anesthetized by using propofol.
  Interventions: Drug: propofol group
- sevoflurane group (Other): The patient who anesthetized by using propofol.
  Interventions: Drug: sevoflurane group

INTERVENTIONS:
Drug: propofol group — Patient will be anesthetized by using propofol infusion during operation
  Other Names: propofol
  Arms: propofol group
Drug: sevoflurane group — Patient will be anesthetized by using sevoflurane inhalation during operation
  Other Names: sevoflurane
  Arms: sevoflurane group

SUMMARY:
Anesthetics agents has variety inflammation during the cancer surgery. This perioperative inflammation can influence to cancer metastasis or recurrence.

The purpose of this study is to prove the variation of immune cell activity between preoperative and postoperative period.

DETAILED DESCRIPTION:
The patients were allocated randomly to receive propofol or sevoflurane. Also, a total of 18ml of blood sample was obtained for total 3 times in consecutive order.

1. immediate before anesthesia induction
2. postoperative 1 hours
3. postoperative 24 hours

Serum in blood will be obtained and activity of helper T cell, natural killer cell and level of serum cytokine will be evaluated by flow cytometry or enzyme-linked immunosorbent assay

ELIGIBILITY:
Inclusion Criteria:

* patient who was planned to undergo colon cancer surgery.

Exclusion Criteria:

* age < 20 years old
* history of hypersensitivity reaction in propofol or sevoflurane
* history of previous cancer
* patient with ongoing inflammation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
natural killer cell activity | preoperative time. postoperative 1 hours and 24 hours
  change of percentage of natural killer cell (scores range from 0 to 100)

SECONDARY OUTCOMES:
helper T cell activity | preoperative time. postoperative 1 hours and 24 hours
  change of percentage of helper T cell (scores range from 0 to 100)

OTHER OUTCOMES:
change of percentage of CD39 and CD73 | preoperative time. postoperative 1 hours and 24 hours
  change of percentage of CD39 and CD73 (scores range from 0 to 100)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D,Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No